CLINICAL TRIAL: NCT03154320
Title: A Trial of Same-Day Testing and Treatment to Improve Outcomes Among Symptomatic Patients Newly Diagnosed With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Weill Medical College of Cornell University (Other); Florida International University (Other); University of California, Davis (Other); Analysis Group, Inc. (Industry)
Responsible Party: Principal Investigator, Serena Patricia Koenig, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI131998
Record Dates: First submitted 2017-03-24; First posted 2017-05-16 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS; Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to standard or same-day treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): On Day 0 (day of HIV diagnosis and study enrollment) participants will receive a chest x-ray and provide a sputum specimen for spot Xpert Ultra testing (48-hour results). Those with high clinical/radiographic suspicion for TB will start same-day TB treatment. On Day 2, participants will return for results of Xpert Ultra testing (spot specimen) and to provide a specimen for early morning Xpert Ultra testing. Those who are Xpert Ultra positive will start TB treatment. Those who are not diagnosed with TB will start ART on Day 7, after testing and treatment for other opportunistic infections. A liquid TB culture will be performed on both the spot and early morning specimens.
  Interventions: Other: Standard treatment
- Same-Day Treatment Group (Experimental): On Day 0 (day of HIV diagnosis and study enrollment) participants will receive a chest x-ray and Xpert Ultra testing with same-day results. Based on clinical symptoms, Xpert Ultra results, and chest x-ray, physician will determine whether or not the participant has tuberculosis. Those who are diagnosed with TB will start same-day TB treatment. Those who are not diagnosed with TB will start same-day ART.
  Interventions: Other: Same-Day Treatment

INTERVENTIONS:
Other: Same-Day Treatment — Treatment with ART or TB medication on day of HIV diagnosis
  Arms: Same-Day Treatment Group
Other: Standard treatment — Standard treatment
  Arms: Standard Group

SUMMARY:
This is a randomized, unblinded study comparing standard vs. same-day treatment for patients with TB symptoms (cough, fever, night sweats, or weight loss) at HIV diagnosis. Six hundred patients will be randomized in a 1:1 ratio to the standard group or the same-day treatment group. All study activities will take place at the GHESKIO Centers in Port-au-Prince, Haiti. The study population includes HIV-infected men and women ≥18 years of age who are ART-naïve, and who present with symptoms of TB (cough, fever, nights sweats, or weight loss) at HIV diagnosis.

DETAILED DESCRIPTION:
This study is a randomized trial that will compare outcomes with standard and same-day treatment among patients with TB symptoms at HIV diagnosis. The standard group will receive same-day chest x-ray as well as Xpert Ultra testing with a spot specimen (with 48-hour turn-around-time). Participants will return for Xpert Ultra results and early morning sputum testing on Day 2. TB treatment will be provided on the day of diagnosis (Day 0 for those with high clinical and radiographic suspicion of TB, and Day 2 for those diagnosed by spot Xpert Ultra). Standard group participants who are not diagnosed with TB will be tested and treated for other opportunistic infections (OIs), as clinically indicated, and will initiate ART on Day 7. The same-day group will receive Xpert Ultra testing (with same-day results) and chest x-ray with same-day ART or TB treatment (on Day 0) based on test results. They will also be tested and treated for other OIs as clinically indicated. They will provide early morning sputum for repeat testing on Day 1. Both groups will receive Xpert Ultra testing on both spot and early morning specimens, with liquid culture on both specimens as the diagnostic gold standard; those with TB will start ART according to WHO guidelines.

Three specific aims are proposed:

Aim 1: To compare the proportion of participants in each group who are alive and in care with undetectable viral load (<200 copies/ml) at 48 weeks after HIV testing. Hypothesis: The proportion of participants retained in care with undetectable viral load will be 51% in the standard and 65% in the same-day group.

Aim 2: To compare mortality in each group at 48 weeks after HIV testing. Hypothesis: Mortality will be 10% in the standard group and 4% in the same-day group.

Aim 3: To conduct a comparison of cost and cost-effectiveness of standard and same-day care, where cost is measured by the mean treatment cost and effectiveness is measured by being alive and in care with plasma HIV-1 RNA level <200 copies/ml at 48 weeks after HIV testing. Hypothesis: Same-day treatment will cost less per patient retained in care with undetectable viral load.

Aim 4: To determine the rates of ART and TB treatment initiation, TB diagnosis after ART initiation, IRIS, adverse events, and adherence in both groups, and to evaluate the sensitivity, specificity, and predictive values of single tests and different testing combinations compared to liquid mycobacterial culture results.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of ≥18 years of age
* Presence of cough, fever, night sweats or weight loss
* Ability and willingness to give written informed consent
* Documentation of positive HIV status (test conducted at GHESKIO)
* Acceptance of HIV diagnosis, defined as affirmative responses to two questions: "I believe that HIV and AIDS exist" and "I believe that the results of my HIV test show that I am infected".

Exclusion Criteria:

* Any use of ART in the past
* Treatment for TB in the year prior to screening visit
* Pregnancy or breastfeeding at the screening visit
* Active drug, alcohol use, or mental condition that would interfere with the ability to adhere to study requirements, in the opinion of the study physician
* Score of <3 for any of the 7 questions on the ART readiness survey
* Planning to transfer care to another clinic during the study period
* Symptoms consistent with WHO stage 4 neurologic disease (cryptococcal meningitis, TB meningitis; central nervous system toxoplasmosis; HIV encephalopathy; progressive multifocal leukoencephalopathy)
* Severe illness, classified as one of the WHO "danger signs" of temperature >39 degrees Celsius, pulse >120 beats/minutes, respiratory rate >30, or inability to walk unaided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Retention in care with viral suppression | 48 weeks after HIV testing
  Proportion of participants who are in care with HIV-1 RNA <200 copies/ml

SECONDARY OUTCOMES:
Mortality | 48 weeks after HIV testing
  All-cause mortality
Mean treatment cost per participant | 48 weeks after HIV testing
  Mean treatment cost per participant
Viral suppression | 48 weeks after HIV testing
  Proportion of participants with HIV-1 RNA <50 copies/ml and <1000 copies/ml
Adherence by medication possession ratio | 48 weeks after HIV testing
  Proportion of participants with 48-week adherence to ART of at least 90% by pharmacy refill records
Adherence by 3-day self-report | 48 weeks after HIV testing
  Proportion of participants with perfect (100%) adherence as measured by 3-day self-report at 48 weeks after HIV testing
Treatment failure | 48 weeks
  Proportion of participants meeting WHO criteria for ART failure and proportion initiating second-line ART during the study period
TB testing characteristics | These diagnostic tests will be conducted during the first week of study enrollment
  Sensitivity, specificity, predictive values, and likelihood ratios of spot and early morning Xpert Ultra results and chest x-ray, as single and as combined tests, with liquid culture as gold standard
Time in clinic | First study day and first study month
  Median time spent in clinic during first day and month of the study
Coping with HIV diagnosis | 2 Weeks, 12 Weeks, 24 Weeks, and 48 Weeks after HIV Testing
  Scores on the COPE survey
Connectedness to Treatment Setting | 2 Weeks, 12 Weeks, 24 Weeks, and 48 Weeks after HIV Testing
  Scores on the Connectedness to Treatment Setting Scale
TB diagnosis after ART initiation | 48-week study period
  Diagnosis of culture-positive TB after ART initiation (BACTEC MGIT 960, Becton Dickinson)
Incidence of immune reconstitution inflammatory syndrome (IRIS) | 48-week study period
  Incidence of paradoxical or unmasking IRIS
Adverse events | 48-week study period
  New Division of AIDS Grade 3 or Grade 4 signs, symptoms, or laboratory abnormalities that are at least a one-grade increase from baseline
Measure of hope and optimism | 2 Weeks, 12 Weeks, 24 Weeks, and 48 Weeks after HIV Testing
  Scores on the State Hope Scale
Patient satisfaction | 12 Weeks, 24 Weeks, and 48 Weeks after HIV Testing
  Scores on the HRSA Patient Satisfaction Survey
Time to death | 48-week study period
  Days to death
Last missed dose of medication | 2 Weeks, 12 Weeks, 24 Weeks, 48 Weeks
  Proportion of participants who report last missed dose of ART was at least 2 weeks ago

CONTACTS AND LOCATIONS:
Overall Officials: Serena P Koenig, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
When the study has been completed, anonymized data will be made publicly available, which will permit replication of reported outcomes.

REFERENCES:
- [Derived] Dorvil N, Rivera VR, Riviere C, Berman R, Severe P, Bang H, Lavoile K, Devieux JG, Faustin M, Saintyl G, Mendicuti MD, Pierre S, Apollon A, Dumond E, Forestal GPL, Rouzier V, Marcelin A, McNairy ML, Walsh KF, Dupnik K, Reif LK, Byrne AL, Bousleiman S, Orvis E, Joseph P, Cremieux PY, Pape JW, Koenig SP. Same-day testing with initiation of antiretroviral therapy or tuberculosis treatment versus standard care for persons presenting with tuberculosis symptoms at HIV diagnosis: A randomized open-label trial from Haiti. PLoS Med. 2023 Jun 9;20(6):e1004246. doi: 10.1371/journal.pmed.1004246. eCollection 2023 Jun. PMID 37294843
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229